CLINICAL TRIAL: NCT02365701
Title: Double-blind, Placebo-controlled, Randomized, 4-week, Phase II Clinical Trial for Assessment of Efficacy and Safety of Motilitone in Patients With Functional Dyspepsia
Brief Title: Study of Motilitone to Treat Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Moti_FD_II
Record Dates: First submitted 2014-09-05; First posted 2015-02-19 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2018-06

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motilitone 30mg (Experimental): Motilitone will be administered in tablet form, 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this medication for 4 weeks.
  Interventions: Drug: Motilitone 30mg
- Placebo (Placebo Comparator): Placebo (same formulation as Motilitone but without the active ingredients) will be administered in tablet form, 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this tablet for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Motilitone 30mg — 30mg of Motilitone in tablet form, to be taken 3 times daily for 4 weeks
  Arms: Motilitone 30mg
Drug: Placebo — Placebo, in tablet form, to be taken 3 times daily for 4 weeks. The placebo is the same formulation as Motilitone except that it does not contain the active pharmaceutical ingredient.
  Arms: Placebo

SUMMARY:
This study is to evaluate efficacy of the investigational drug Motilitone at 90 mg in patients with Functional Dyspepsia as measured by change in maximum tolerated volume and aggregate symptom score on the nutrient drink test.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subject fulfilling Rome III criteria for Functional Dyspepsia: They must have one or more of the following:

  1. Bothersome postprandial fullness
  2. Early satiation
  3. Epigastric pain
  4. Epigastric burning AND No evidence of structural disease at upper endoscopy within last 3 months that is likely to explain the symptoms These must be fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
* (2) At least a moderate or severe level within the previous 3 months for two of the following eight symptoms: upper abdominal pain, upper abdominal discomfort, postprandial fullness, upper abdominal bloating, early satiation, nausea, vomiting or excessive belching (each symptom rated as 0: None, 1: Mild, 2: Moderate, 3: Severe).
* (3) Subjects should be able to provide a written informed consent.

Exclusion Criteria:

* (1) Subject currently on medication for another study or who participated in another clinical trial or study within 4 weeks before the start of this study.
* (2) Women of childbearing potential who are not using contraception and pregnant or lactating women.
* (3) Subject who had surgery that may affect gastrointestinal motility.
* (4) Subject with known history of gastric bleeding, intestinal obstruction or perforation.
* (5) Subject with known history of celiac disease, inflammatory bowel disease (Crohn's disease, ulcerative colitis) or microscopic colitis.
* (6) Subject who had any of the diseases such as reflux esophagitis, gastroduodenal ulcer, gastric adenocarcinoma, esophageal adenocarcinoma, pancreatic disease, etc. that may be an organic cause of dyspepsia.
* (7) Subject with liver dysfunction (serum glutamic oxaloacetic transaminase/serum glutamic pyruvic transaminase is at least 2.5 times higher than ULN).
* (8) Subject with renal dysfunction (Serum creatinine level is at least 1.5 times higher than ULN).
* (9) Subject with a serious cardiovascular (including known baseline QT prolongation defined by >450 msec) or respiratory illness.
* (10) Subject with diagnosed psychotic illnesses, substance dependence or alcoholism.
* (11) Subject currently taking drugs that may affect gastrointestinal motility (e.g., anticholinergic, Reglan, erythromycin, azithromycin, Domperidone, etc.), Buspirone, Acotiamide, Tramadol, nonsteroidal anti-inflammatory drug, systemic corticosteroids, and antidepressants, etc. within last 2 weeks of randomization.
* (12) Medications that can affect QT within last 2 weeks of randomization.
* (13) Subjects on herbal supplements for Functional Dyspepsia within last 2 weeks of randomization.
* (14) Subjects with gastric electric stimulator in place.
* (15) Subjects on narcotics or benzodiazepines within 7 days of randomization.
* (16) Subjects with score > 12 for anxiety or depression on the Hospital Anxiety and Depression Scale (HADS).
* (17) Vulnerable study population

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in maximum tolerated volume by nutrient drink test | week -2, week 4
Change in aggregate symptom score by nutrient drink test | week -2, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States